CLINICAL TRIAL: NCT02899078
Title: Phase Ib/II Trial of Ibrutinib Plus Nivolumab in Patients With Previously-Treated Metastatic Renal Cell Cancer
Brief Title: Ibrutinib and Nivolumab in Treating Patients With Previously-Treated Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 895892; UCDCC#262 (Registry Identifier: UC Davis); UCDCC#262 (Other: University of California Davis Comprehensive Cancer Center); NCI-2016-01266 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-08-30; First posted 2016-09-14 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ibrutinib, nivolumab) (Experimental): Patients receive ibrutinib PO QD on days 1-28 and nivolumab intravenously IV over 60 minutes on days 1 and 15. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; IMBRUVICA
Drug: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; Opdivo; NIVO

SUMMARY:
This phase Ib/II trial studies how well ibrutinib and nivolumab work in treating patients with previously-treated kidney cancer that has spread to other parts of the body. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving Ibrutinib and nivolumab may work better in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess in a preliminary fashion the feasibility and efficacy of ibrutinib in combination with nivolumab in patients with previously-treated metastatic renal cell cancer (mRCC).

SECONDARY OBJECTIVE:

To evaluate the safety of the combination of ibrutinib and nivolumab in patients with previously treated mRCC.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell cancer patients (any histologic subtype) with measurable and/or evaluable disease who have completed at least one line of prior systemic therapy are potentially eligible for this trial; any number of prior systemic therapies are allowed, including prior nivolumab
* Absolute neutrophil count > 750 cells/mm^3 (0.75 x 10^9/L)
* Platelet count > 50,000 cells/mm^3 (50 x 10^9/L)
* Hemoglobin > 8.0 g/dL
* Serum aspartate transaminase (aspartate aminotransferase [AST]) or alanine transaminase (alanine aminotransferase [ALT]) =< 3.0 x upper limit of normal (ULN)
* Estimated creatinine clearance >= 30 ml/min (Cockcroft-Gault)
* Bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative serum pregnancy test upon study entry
* Male and female subjects who agree to use both a highly effective methods of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) and a barrier method (e.g., condoms, cervical ring, sponge, etc.) during the period of therapy and for 30 days after the last dose of study drug

Exclusion Criteria:

* Cytotoxic chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 4 weeks prior to first administration of study treatment and/or other renal cell carcinoma (RCC)-directed systemic therapy =< 2 weeks prior to first administration of study treatment
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease
  * Adequately treated carcinoma in situ or T1 urothelial cancer without evidence of disease
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration [> 14 days] of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent infection requiring systemic treatment that was completed =< 14 days before the first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* Any uncontrolled active systemic infection
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, known autoimmune disease, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Concomitant use of warfarin or other vitamin K antagonists; Note: Subjects receiving antiplatelet agents in conjunction with ibrutinib should be observed closely for any signs of bleeding or bruising, and ibrutinib should be withheld in the event of any bleeding events; supplements such as fish oil and vitamin E preparations should be avoided
* Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* QT prolongation and/or familiar history of QT prolongation and uncontrolled cardiac arrhythmias
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo Lara, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ibrutinib, Nivolumab): Patients receive ibrutinib PO QD on days 1-28 and nivolumab intravenously IV over 60 minutes on days 1 and 15. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Ibrutinib: Given PO Nivolumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Started | 31
Completed | 28
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From baseline to death or progression, assessed for up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Number analyzed (Participants) | 28
months | 2.5 [1.9 to 4.8]

2. Secondary Outcome: National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03
Description: Number of participants with adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
Time Frame: Up to 30 days
Measure: Number; unit: participants
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Number analyzed (Participants) | 31
participants | 31

3. Secondary Outcome: Overall Survival
Description: Overall survival, calculated using the Kaplan-Meier method as the duration from start of treatment to death by any cause.
Time Frame: Up to 32 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Number analyzed (Participants) | 28
months | 9.1 [6.6 to 19.0]

4. Secondary Outcome: Response
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Treatment (Ibrutinib, Nivolumab)
Number analyzed (Participants) | 28
percentage of evaluable participants | 10.7 [3.7 to 27.2]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from enrollment until 30 days after last dose of study drug. All-Cause Mortality was from first dose until death, assessed up to about 28 months.
Description: Incidence of adverse events according to CTCAE v4.0
Arm/Group | Treatment (Ibrutinib, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 16/31
Serious Adverse Events (participants affected / at risk) | 17/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment (Ibrutinib, Nivolumab) (N=31)
Urinary tract infection (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1/1
Gastric hemorrhage (Gastrointestinal disorders) | 1/1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1/1
Nausea (Gastrointestinal disorders) | 1/1
Vomiting (Gastrointestinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ibrutinib, Nivolumab) (N=31)
Anemia (Blood and lymphatic system disorders) | 11
Lymphocyte count reduction (Investigations) | 12
Fatigue (General disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT02899078/Prot_SAP_000.pdf